CLINICAL TRIAL: NCT03390192
Title: Investigation for Individualized Noninvasive Neuromodulation in Neurorehabilitation of Brain Disease: Longitudinal Study
Brief Title: Noninvasive Dual-mode Stimulation Therapy for Neurorehabilitation in Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2013-06-002-009
Record Dates: First submitted 2017-12-25; First posted 2018-01-04 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2017-12

CONDITIONS: Stroke
Keywords: Noninvasive brain stimulation; Repetitive Transcranial Magnetic Stimulation; Transcranial Direct Current Stimulation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Device: No

ARMS (2):
- Dual-mode stimulation (Experimental): Dual-mode stimulation is applied over the bilateral primary motor cortex (M1) using active rTMS and active tDCS. 1 Hz of rTMS is applied over the contralesional M1 for 20 minutes with simultaneous application of anodal tDCS on the ipsilesional M1.
  Each participant's total FMA score is assessed and their resting-state fMRI data at two times: prior to stimulation (pre-stimulation) and 2 months after stimulation (post-stimulation) are acquired.
  Interventions: Device: Dual-mode stimulation
- Single sham stimulation (Active Comparator): Single sham stimulation is applied over the bilateral primary motor cortex (M1) using active rTMS and sham tDCS. 1 Hz of rTMS over the contralesional M1 was applied for 20 minutes with simultaneous application of tDCS with sham mode (no stimulation) on the ipsilesional M1.
  Each participant's total FMA score is assessed and their resting-state fMRI data at two times: prior to stimulation (pre-stimulation) and 2 months after stimulation (post-stimulation) are acquired.
  Interventions: Device: Single sham stimulation

INTERVENTIONS:
Device: Dual-mode stimulation — 1Hz rTMS over contralesional primary motor cortex and anodal tDCS over ipsilesional primary motor cortex are simultaneously simulated.
  Arms: Dual-mode stimulation
Device: Single sham stimulation — 1Hz rTMS over contralesional primary motor cortex and sham tDCS (no stimulation) over ipsilesional primary motor cortex are simultaneously simulated.
  Arms: Single sham stimulation

SUMMARY:
Repetitive transcranial magnetic stimulation (rTMS) or transcranial direct current stimulation (tDCS) has been used for the modulation of stroke patients' motor function by altering the cortical excitability. Recently, more challenging approaches, such as stimulation of two or more sites or use of dual modality have been studied in stroke patients. In this study, simultaneous stimulation using both inhibitory rTMS (1Hz) and anodal tDCS (dual-mode stimulation) over bilateral primary motor cortices (M1s) was investigated to compare its modulatory effects with single inhibitory rTMS stimulation in subacute stroke patients.

ELIGIBILITY:
Inclusion Criteria:

* First-ever stroke patients
* Subacute stage (less than 4 weeks)
* Total Fugl-Meyer Assessment (FMA) score under 84

Exclusion Criteria:

* Major active neurological disease or psychiatric disease
* A history of seizure
* Metallic implants in their brain

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2015-01-13 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment score | 2 months post-stimulation
  Fugl-Meyer Assessment score reflects a motor impairment of a patient. Score range is between 0 and 100.

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee J, Lee A, Kim H, Shin M, Yun SM, Jung Y, Chang WH, Kim YH. Different Brain Connectivity between Responders and Nonresponders to Dual-Mode Noninvasive Brain Stimulation over Bilateral Primary Motor Cortices in Stroke Patients. Neural Plast. 2019 Apr 7;2019:3826495. doi: 10.1155/2019/3826495. eCollection 2019. PMID 31093270